CLINICAL TRIAL: NCT04101162
Title: Diagnostic Accuracy in a New Ultrasound Software Compared to Histology for Non Alcoholic Fatty Liver Disease (NAFLD) and Non Alcoholic Steato Hepatitis (NASH) in Morbidly Obese Individuals Undergoing Bariatic Surgery and/or Cholecystectomy
Brief Title: NAFLD Study: US vs Liver Biopsy
Acronym: NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0109926/2018
Record Dates: First submitted 2019-09-05; First posted 2019-09-24 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liver biopsy (Other)
  Interventions: Diagnostic Test: shear waves elastography; liver biopsy
- ATI (Other)
  Interventions: Diagnostic Test: shear waves elastography; liver biopsy

INTERVENTIONS:
Diagnostic Test: shear waves elastography; liver biopsy — Diagnostic accuracy in a new ultrasound software compared to histology for Non Alcoholic Fatty liver disease (NAFLD) and Non Alcoholic Steato Hepatitis (NASH)

SUMMARY:
Evaluate the diagnostic accuracy of the new ultrasound software vs hepatic histology, the current reference standard for the diagnosis of NAFLD and NASH in 20 obese patients (BMI> 30) candidates for laparoscopic bariatric surgery and / or cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are candidates for bariatric surgery between the ages of 18 and 65,

   * BMI> 40 kg / m2, in the absence of any other comorbidity
   * BMI> 35 kg / m2, in the presence of comorbidities among those classically considered to be associated with obesity
   * ICM> 30 kg / m2, in the presence of T2DM not in glycometabolic compensation
2. Patients who are candidates for laparoscopic cholecystectomy for symptomatic calculi with BMI> 30

Exclusion Criteria:

* Age ≤ 18 or ≥ 65
* Any concurrent surgical procedure except cholecystectomy and hiatal hernia repair
* Conversion into laparotomy surgery
* Post-operative complications requiring new surgical treatment
* Patient not compliant in the follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
diagnostic accurancy of ATI in obese patients | 6 months
  a new ultrasound software compared with liver biopsy in obese patients.

CONTACTS AND LOCATIONS:
Locations (1):
- ICOT Latina, Latina, LT, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT04101162/Prot_000.pdf